CLINICAL TRIAL: NCT00854815
Title: Irrigation Versus No Irrigation for Perforated Appendicitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Principal Investigator, Shawn St. Peter, MD, Children's Mercy Hospital Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08 11 181
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Perforated Appendicitis
Keywords: Perforated appendicitis; laparoscopic appendectomy; children; irrigation
MeSH Terms: conditions — Appendicitis | interventions — Therapeutic Irrigation; WASH protein, Drosophila; Suction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Irrigation (Active Comparator): Irrigation of the area with at least 500ml normal saline using the power suction/irrigator
  Interventions: Procedure: Irrigation
- No Irrigation (Active Comparator): Only suction with the power suction/irrigator without saline attached
  Interventions: Procedure: No Irrigation

INTERVENTIONS:
Procedure: Irrigation — Irrigation of the area with at least 500ml NS using the power suction/irrigator
  Other Names: washout
  Arms: Irrigation
Procedure: No Irrigation — Suction only using suction/irrigator
  Other Names: suction
  Arms: No Irrigation

SUMMARY:
The purpose is to quantify the effect of irrigation during laparoscopic appendectomy for perforated appendicitis.

DETAILED DESCRIPTION:
This will be a prospective, randomized clinical trial involving patients who present to the hospital with perforated appendicitis. This will be a definitive study.

Power calculation was based on abscess rate in the previous prospective study. An unacceptable abscess rate needed to be chosen. Our current rate is 20%, or one-fifth of the patients. If this were to increase by 15%, it would place just over one third of the patients at risk which would be unacceptable. This is comparable to the 36% rejection level we used for the previous IRB approved trial (#07 02-031). Using a delta of 0.15 with alpha of 0.05 and power of 0.8, the sample size is 109 patients in each arm. Therefore we will anticipate enrolling 220.

Subjects will be those children who are found to have severe inflammatory changes on imaging or a high clinical suspicion of perforation. Permission will be obtained from parents prior to the operation. All of these children will be under duress prior to randomization, therefore we request waiving assent as we have done with the previous perforated appendicitis studies.

The final decision to include a child in the study will made after perforation has been visually confirmed during surgery. Perforation will be defined as an identifiable hole in the appendix or stool in the abdomen. The randomization assignment will be made known at the initiation of the operation, and confirmation of perforation will confirm the patient will utilize the next randomization slot.

The irrigation group will have suction irrigator set up with a 1 liter bag of normal saline. The surgeon must use at least 500 ml of this bag but may use as much as they choose.

The no irrigation group will have the suction irrigator set up without the saline attachment. This will leave them with the capacity for suction only. Since several suction devices exist, this will assure the same type of suction for both groups.

After the operation, both groups will be managed in the same manner. When the patient is tolerating a regular diet, on oral pain medication and has been afebrile for over 12 hours, they will be discharged on oral antibiotics to complete a course of 7 days. If they stay until the 5th post-operative day, a white blood cell count will be checked, which if it is normal, they will be discharged to home without antibiotics. This is standard post-operative care as delineated by our previous prospective, randomized.

ELIGIBILITY:
Inclusion Criteria:

* Under 18 yrs old
* Perforation identified as hole in the appendix or fecalith in the abdomen

Exclusion Criteria:

* No perforation
* A significant comorbidity that would limit their ability to recover from appendectomy in a normal fashion

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Estimated)
Dates: Start 2008-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Post-operative abscess | 1 month

SECONDARY OUTCOMES:
operating time | 1 day
length of stay | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shawn D St. Peter, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States